CLINICAL TRIAL: NCT01082445
Title: Effects of Prolonged N-acetylcysteine Administration on Foot Ulcer Oxygenation in Diabetic Patients
Brief Title: Effects of N-acetylcysteine on Diabetic Foot Oxygenation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Valentino Martina, Aggregated Professor, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NACPIEDE
Record Dates: First submitted 2010-03-04; First posted 2010-03-08 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Foot Ulcer, Diabetic
Keywords: stage C; grade 0 (Texas University)
MeSH Terms: conditions — Diabetic Foot | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-acetylcysteine (Experimental): 50 patients that receive 600 mg of acetylcysteine for 3 times a day.
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): 50 subjects taking placebo pills 3 times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — 600 mg, 1 tablet 3 times a day for 3 months
  Other Names: Fluimucil (R) 600 mg, tablets
  Arms: N-acetylcysteine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether N-acetylcysteine is effective in the treatment or prevention of the foot ulcers in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 70 years.
* Type 1 or 2 diabetes mellitus with foot ulcer (grade 0 stage C according to Texas University Classification).
* Written informed consent.

Exclusion Criteria:

* N-acetylcysteine assumption in the 6 months previous to the study.
* Hypersensibility to acetylcysteine.
* Neoplasms, severe systemic, hepatic, pulmonary, cardiovascular or renal diseases.
* Psychiatric diseases or drug abuse problems.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Tissue oxygenation improvement | Basal (time 0) and after 3 months of treatment/observation

SECONDARY OUTCOMES:
Improvement of the endothelial function | Basal (time 0) and after 3 months of treatment/observation
  nitrites/nitrates - ICAM - VCAM - PAI-1
Oxidation status reduction | Basal (time 0) and after 3 months of treatment/observation
  8-iso PGF-2alpha assessment

CONTACTS AND LOCATIONS:
Overall Officials: Valentino Martina, Professor, Principal Investigator — University of Turin, Italy
Locations (1):
- Div. Endocrinology, Diabetology and Metabolism - University of Turin, Turin, TO, Italy

REFERENCES:
- [Background] Martina V, Masha A, Gigliardi VR, Brocato L, Manzato E, Berchio A, Massarenti P, Settanni F, Della Casa L, Bergamini S, Iannone A. Long-term N-acetylcysteine and L-arginine administration reduces endothelial activation and systolic blood pressure in hypertensive patients with type 2 diabetes. Diabetes Care. 2008 May;31(5):940-4. doi: 10.2337/dc07-2251. Epub 2008 Feb 11. PMID 18268065
- [Background] Masha A, Brocato L, Dinatale S, Mascia C, Biasi F, Martina V. N-acetylcysteine is able to reduce the oxidation status and the endothelial activation after a high-glucose content meal in patients with Type 2 diabetes mellitus. J Endocrinol Invest. 2009 Apr;32(4):352-6. doi: 10.1007/BF03345726. PMID 19636205
- [Background] Martina V, Bruno GA, Zumpano E, Origlia C, Quaranta L, Pescarmona GP. Administration of glutathione in patients with type 2 diabetes mellitus increases the platelet constitutive nitric oxide synthase activity and reduces PAI-1. J Endocrinol Invest. 2001 Jan;24(1):37-41. doi: 10.1007/BF03343806. PMID 11227730
- [Background] Ignarro LJ, Edwards JC, Gruetter DY, Barry BK, Gruetter CA. Possible involvement of S-nitrosothiols in the activation of guanylate cyclase by nitroso compounds. FEBS Lett. 1980 Feb 11;110(2):275-8. doi: 10.1016/0014-5793(80)80091-3. No abstract available. PMID 6102928
- See also: International Working Group on the Diabetic Foot — http://www.iwgdf.org/